CLINICAL TRIAL: NCT04578288
Title: Individualized Blood Pressure Management During Endovascular Treatment of Acute Ischemic Stroke Under Procedural Sedation
Brief Title: Individualized Blood Pressure Management During Endovascular Stroke Treatment
Acronym: INDIVIDUATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. Silvia Schönenberger, MD, Principal Investigator, Co-principal investigator: Dr. Min Chen, MD, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Heidelberg University Hospital
Record Dates: First submitted 2020-09-09; First posted 2020-10-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Blood Pressure management (Active Comparator): The standard blood pressure management is maintenance of intraprocedural pre-recanalization SBP between 140-180 mmHg for all patients who receive endovascular thrombectomy for acute ischemic stroke in anterior circulation.
  Interventions: Procedure: INDIVIDUALIZED BLOOD PRESSURE MANAGEMENT DURING ENDOVASCULAR TREATMENT OF ACUTE ISCHEMIC STROKE UNDER PROCEDURAL SEDATION
- Individualized Blood Pressure management (Experimental): The study intervention would be maintaining the intraprocedural pre-recanalization blood pressure in individualized SBP target ranges depending on the systolic blood pressure of the patient at presentation (=baseline SBP or bSBP).
  Interventions: Procedure: INDIVIDUALIZED BLOOD PRESSURE MANAGEMENT DURING ENDOVASCULAR TREATMENT OF ACUTE ISCHEMIC STROKE UNDER PROCEDURAL SEDATION

INTERVENTIONS:
Procedure: INDIVIDUALIZED BLOOD PRESSURE MANAGEMENT DURING ENDOVASCULAR TREATMENT OF ACUTE ISCHEMIC STROKE UNDER PROCEDURAL SEDATION — The individual target range is defined as: bSBP ± 10 mmHg. The lowest possible SBP target range is 100-120 mmHg. The highest SBP target range is determined on the basis of whether patients receive concurrent IV fibrinolytic therapy or not. In patients where IV fibrinolytic therapy is applied, the highest SBP range is 160-180 mmHg, in patients without concurrent fibrinolytic therapy the highest SBP range is 180-200 mmHg.

SUMMARY:
Optimal blood pressure management during endovascular treatment of acute ischemic stroke is not well established. Several retrospective data indicate, that there is a U-shaped relationship of admission blood pressure and functional outcome, where either very high or very low blood pressure are disadvantageous for the patient. Low blood pressure might lead to hypoperfusion in ischemic areas (i.e. penumbra) and to larger infarction sizes, while on the other hand, maladaptive high blood pressure might lead to edema and hemorrhage. Retrospective data investigating intraprocedural blood pressure and its influence on outcome is limited. Some studies indicate that hypotensive blood pressure drops from the level of the admission blood pressure lead to a worse outcome. Intraprocedural hypotensive drops are common during endovascular thrombectomy due to application of necessary sedative drugs for agitated stroke patients. We aim to investigate whether individualized blood pressure management with patient-specific blood pressure targets situated at the level during presentation might be associated with better functional outcome compared with general blood pressure targets for patients during thrombectomy. For this purpose, we plan to perform this single center, parallel-group, open-label randomized controlled trial with blinded endpoint evaluation (PROBE).

ELIGIBILITY:
Inclusion Criteria:

1. Decision for thrombectomy according to local protocol for acute recanalizing stroke treatment
2. Age 18 years or older, either sex
3. National Institutes of Health Stroke Scale (NIHSS) ≥ 8
4. Acute ischemic stroke in the anterior circulation with isolated or combined occlusion of: Internal carotid artery (ICA) and/or middle cerebral artery (MCA)
5. Informed consent by the patient him-/herself or his/her legal representative obtainable within 72 h of treatment

Exclusion Criteria:

1. Intracerebral hemorrhage
2. Coma on admission (Glasgow Coma Scale ≤ 8)
3. Severe respiratory instability, loss of airway protective reflexes or vomiting on admission, where primary intubation and general anesthesia is deemed necessary
4. Intubated state before randomization
5. Severe hemodynamic instability (e.g. due to decompensated heart insufficiency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Functional outcome 90 days after stroke onset | 90 days
  modified Rankin scale (mRS) after 90 days dichotomized 0-2 by (favorable outcome) to 3-6 (unfavorable outcome).

SECONDARY OUTCOMES:
Early neurological improvement indicated by change of National Institute of Health Stroke Scale (NIHSS) Score 24 hours after admission | 24 hours
  [NIHSS on admission - NIHSS after 24 hours]
Infarction size, determined with MRI or (in case of contraindications CT scan) 12-36 h after admission on a post-interventional follow up scan [milliliter] | 12-36 hours
  Infarction size 12-36 hours after symptom onset
Time of intraprocedural SBP in target range [percentage of time in target range between groin puncture and reperfusion] | Duration of thrombectomy procedure up to 240 minutes
  Duration of thrombectomy procedure
Time of intraprocedural SBP spent in treatment range ± 10 mmHg [percentage of time in range between groin puncture and reperfusion] | Duration of thrombectomy procedure up to 240 minutes
  Duration of thrombectomy procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rasmussen M, Schonenberger S, Henden PL, Valentin JB, Espelund US, Sorensen LH, Juul N, Uhlmann L, Johnsen SP, Rentzos A, Bosel J, Simonsen CZ; SAGA collaborators. Blood Pressure Thresholds and Neurologic Outcomes After Endovascular Therapy for Acute Ischemic Stroke: An Analysis of Individual Patient Data From 3 Randomized Clinical Trials. JAMA Neurol. 2020 May 1;77(5):622-631. doi: 10.1001/jamaneurol.2019.4838. PMID 31985746
- [Background] Lowhagen Henden P, Rentzos A, Karlsson JE, Rosengren L, Sundeman H, Reinsfelt B, Ricksten SE. Hypotension During Endovascular Treatment of Ischemic Stroke Is a Risk Factor for Poor Neurological Outcome. Stroke. 2015 Sep;46(9):2678-80. doi: 10.1161/STROKEAHA.115.009808. Epub 2015 Jul 14. PMID 26173727
- [Background] Schonenberger S, Uhlmann L, Ungerer M, Pfaff J, Nagel S, Klose C, Bendszus M, Wick W, Ringleb PA, Kieser M, Mohlenbruch MA, Bosel J. Association of Blood Pressure With Short- and Long-Term Functional Outcome After Stroke Thrombectomy: Post Hoc Analysis of the SIESTA Trial. Stroke. 2018 Jun;49(6):1451-1456. doi: 10.1161/STROKEAHA.117.019709. Epub 2018 May 2. PMID 29720440
- [Background] Whalin MK, Halenda KM, Haussen DC, Rebello LC, Frankel MR, Gershon RY, Nogueira RG. Even Small Decreases in Blood Pressure during Conscious Sedation Affect Clinical Outcome after Stroke Thrombectomy: An Analysis of Hemodynamic Thresholds. AJNR Am J Neuroradiol. 2017 Feb;38(2):294-298. doi: 10.3174/ajnr.A4992. Epub 2016 Nov 3. PMID 27811133
- [Background] Petersen NH, Ortega-Gutierrez S, Wang A, Lopez GV, Strander S, Kodali S, Silverman A, Zheng-Lin B, Dandapat S, Sansing LH, Schindler JL, Falcone GJ, Gilmore EJ, Amin H, Cord B, Hebert RM, Matouk C, Sheth KN. Decreases in Blood Pressure During Thrombectomy Are Associated With Larger Infarct Volumes and Worse Functional Outcome. Stroke. 2019 Jul;50(7):1797-1804. doi: 10.1161/STROKEAHA.118.024286. Epub 2019 Jun 4. PMID 31159701
- [Derived] Chen M, Sauer LD, Potreck A, Kieser M, Bendszus M, Ringleb P, Mohlenbruch M, Schonenberger S. Association of hemodynamic variability during endovascular stroke treatment with functional outcome and parenchymal hemorrhage. Ther Adv Neurol Disord. 2025 Nov 24;18:17562864251391837. doi: 10.1177/17562864251391837. eCollection 2025. PMID 41306441
- [Derived] Chen M, Meis J, Potreck A, Sauer LD, Kieser M, Bendszus M, Wick W, Ringleb PA, Mohlenbruch MA, Schonenberger S. Effect of Individualized Versus Standardized Blood Pressure Management During Endovascular Stroke Treatment on Clinical Outcome: A Randomized Clinical Trial. Stroke. 2023 Nov;54(11):2755-2765. doi: 10.1161/STROKEAHA.123.044062. Epub 2023 Sep 21. PMID 37732489
- [Derived] Chen M, Kronsteiner D, Mohlenbruch MA, Kieser M, Bendszus M, Wick W, Nagel S, Ringleb PA, Schonenberger S. Individualized blood pressure management during endovascular treatment of acute ischemic stroke under procedural sedation (INDIVIDUATE) - An explorative randomized controlled trial. Eur Stroke J. 2021 Sep;6(3):276-282. doi: 10.1177/23969873211000879. Epub 2021 Mar 4. PMID 34746424